CLINICAL TRIAL: NCT04768205
Title: The Efficacy of Kinesio Taping With Therapy in the Treatment of Globus Pharyngeus: a Randomized Sham-controlled Trial
Brief Title: The Efficacy of Kinesio Taping With Therapy in the Treatment of Globus Pharyngeus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Yavuz Atar, Associate Professor, M.D., Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 60
Record Dates: First submitted 2021-02-20; First posted 2021-02-24 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Globus Pharyngeus
Keywords: kinesio taping; globus; globus pharyngeus; sensation; therapy
MeSH Terms: conditions — Globus Sensation | interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Study group (Active Comparator): The therapy and Kinesio tex gold tape that was affixed to stretched and neck localised were applied
  Interventions: Device: Kinesio tape
- Sham control group (Placebo Comparator): The therapy and Kinesio tex gold tape that was affixed to different neck localised as no-stretched were applied
  Interventions: Device: Kinesio tape

INTERVENTIONS:
Device: Kinesio tape — The Kinesio tex tape is a medical tape that had been certified and patented.

SUMMARY:
Globus pharyngeus or sensation may be defined as a feeling of something a lump in the throat without dysphagia. Kinesio tex tape is a medical tap developed by Dr. Kase for therapeutic purposes and has been widely used in physical therapy applications in recent years. Although it is not a treatment with full consensus, the patient's complaints can be corrected with a small number of different therapy techniques or regulations on life.

DETAILED DESCRIPTION:
We conducted a therapy program with kinesio taping on patients who diagnosed with globus pharyngeus for 8 session with sham kinesio taping controlled group. This study aimed to assess of efficacy of the kinesio taping with therapy on patients patients who diagnosed with globus pharyngeus.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with globus pharyngeus
* 18 -65 years
* give a consent form

Exclusion Criteria:

* patients with dysphagia or odynophagia
* laryngeal organic pathologies
* pharyngeal organic pathologies
* epiglottic retroversion
* malignancy
* pregnancy
* mental disorders
* neurological disorders
* major psychiatric disorders
* give not a consent form

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-08-30 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
The outcomes of Glasgow Edinburg Throat Scale | Baseline
  It was assessed by Turkish validated Glasgow Edinburg Throat Scale that a self questionnaire in globus pharyngeus patients. The minimum score is 0 and maximum score is 7 per question. The high scores were worst low scores were good.
The outcomes of Glasgow Edinburg Throat Scale | 4 weeks
  It was assessed by Turkish validated Glasgow Edinburg Throat Scale that a self questionnaire in globus pharyngeus patients. The minimum score is 0 and maximum score is 7 per question. The high scores were worst low scores were good.
The outcomes of Glasgow Edinburg Throat Scale | 2 months
  It was assessed by Turkish validated Glasgow Edinburg Throat Scale that a self questionnaire in globus pharyngeus patients. The minimum score is 0 and maximum score is 7 per question. The high scores were worst low scores were good.
The outcomes of Beck depression inventory | Baseline
  It was assessed by Turkish validated depression inventory that a questionnaire about psychosocial situations. The minimum score is 0 and maximum score is 3 per question. The high scores were worst low scores were good.
The outcomes of Beck depression inventory | 4 weeks
  It was assessed by Turkish validated Beck depression inventory that a questionnaire about psychosocial situations. The minimum score is 0 and maximum score is 3 per question. The high scores were worst low scores were good.
The outcomes of Beck depression inventory | 2 months
  It was assessed by Turkish validated Beck depression inventory that a questionnaire about psychosocial situations. The minimum score is 0 and maximum score is 3 per question. The high scores were worst low scores were good.
The outcomes of Beck anxiety inventory | Baseline
  It was assessed by Turkish validated Beck anxiety inventory that a questionnaire about psychosocial situations. The minimum score is 0 and maximum score is 3 per question. The high scores were worst low scores were good.
The outcomes of Beck anxiety inventory | 4 weeks
  It was assessed by Turkish validated Beck anxiety inventory that a questionnaire about psychosocial situations. The minimum score is 0 and maximum score is 3 per question. The high scores were worst low scores were good.
The outcomes of Beck anxiety inventory | 2 months
  It was assessed by Beck anxiety inventory that a questionnaire about psychosocial situations. The minimum score is 0 and maximum score is 3 per question. The high scores were worst low scores were good.
The visual analog scale | Baseline
  The globus sense was assessed by visual analog scale. The minimum score is 0 and maximum score is 100 on a line as 100 millimetres . The high scores were worst low scores were good.
The visual analog scale | 4 weeks
  The globus sense was assessed by visual analog scale. The minimum score is 0 and maximum score is 100 on a line as 100 millimetres. The high scores were worst low scores were good.
The visual analog scale | 2 months
  The globus sense was assessed by visual analog scale. The minimum score is 0 and maximum score is 100 on a line as 100 millimetres. The high scores were worst low scores were good.

SECONDARY OUTCOMES:
Eating Assessment Tool | Baseline
  The Turkish validated questionnaire consists of 10 questions that scores are from 0 to 40. Low score is better, higher score is worse.
Eating Assessment Tool | 4 weeks
  The Turkish validated questionnaire consists of 10 questions that scores are from 0 to 40. Low score is better, higher score is worse.
Eating Assessment Tool | 2 months
  The Turkish validated questionnaire consists of 10 questions that scores are from 0 to 40. Low score is better, higher score is worse.
The outcomes of voice handicap index - 10 | Baseline
  It was assessed by Turkish validated voice handicap index - 10 that a self questionnaire in patients. The minimum score is 0 and maximum score is 4 per question. The high scores were worst low scores were good.
The outcomes of voice handicap index - 10 | 4 weeks
  It was assessed by Turkish validated voice handicap index - 10 that a self questionnaire in patients. The minimum score is 0 and maximum score is 4 per question. The high scores were worst low scores were good.
The outcomes of voice handicap index - 10 | 2 months
  It was assessed by Turkish validated voice handicap index - 10 that a self questionnaire in patients. The minimum score is 0 and maximum score is 4 per question. The high scores were worst low scores were good.
The outcomes of reflux symptom index | Baseline
  The laryngopharyngeal reflux was assessed by Turkish validated reflux symptom index - 10 that a self questionnaire in patients. The minimum score is 0 and maximum score is 5 per question. The high scores were worst low scores were good.
The outcomes of reflux symptom index | 4 weeks
  The laryngopharyngeal reflux was assessed by Turkish validated reflux symptom index - 10 that a self questionnaire in patients. The minimum score is 0 and maximum score is 5 per question. The high scores were worst low scores were good.
The outcomes of reflux symptom index | 2 months
  The laryngopharyngeal reflux was assessed by Turkish validated reflux symptom index - 10 that a self questionnaire in patients. The minimum score is 0 and maximum score is 5 per question. The high scores were worst low scores were good.
Penetration and aspiration scale | Baseline
  The scale consists of 8 levels for assessment of penetration and aspiration. The scores are from 0 to 8. Low score is better, higher score is worse.
Yale pharyngeal residue severity rating scale | Baseline
  The scale consists of 5 assessment units for pharyngeal residue. The scores are from 1 to 5. Low score is better, higher score is worse.

OTHER OUTCOMES:
Subject demographics | Baseline
  The median values of age and ratio of gender in all groups

CONTACTS AND LOCATIONS:
Overall Officials: Yavuz Atar, Asso Prof,MD, Study Chair — University of Health Sciences, ENT Clinic, Prof Dr Cemil Tascioglu City Hospital; Sevgi Atar, MD, Study Director — University of Health Sciences, PMR Clinic, Prof Dr Cemil Tascioglu City Hospital
Locations (1):
- Prof Dr Cemil Tascioglu City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khalil HS, Bridger MW, Hilton-Pierce M, Vincent J. The use of speech therapy in the treatment of globus pharyngeus patients. A randomised controlled trial. Rev Laryngol Otol Rhinol (Bord). 2003;124(3):187-90. PMID 14725135
- [Background] Morris D, Jones D, Ryan H, Ryan CG. The clinical effects of Kinesio(R) Tex taping: A systematic review. Physiother Theory Pract. 2013 May;29(4):259-70. doi: 10.3109/09593985.2012.731675. Epub 2012 Oct 22. PMID 23088702